CLINICAL TRIAL: NCT06392568
Title: Epidemiological Features of Emergent Highly Resistant Bacteria in Tunisian Intensive Care Units: A Prospective Multicenter National Observational Study (NOSOREA-3)
Brief Title: Epidemiological Features of Emergent Highly Resistant Bacteria in Tunisian Intensive Care Units
Acronym: NOSOREA3
Status: Recruiting | Type: Observational
Sponsor: Abderrahmane Mami Hospital (Other)
Responsible Party: Principal Investigator, Amira JAMOUSSI, Professor, Abderrahmane Mami Hospital
Other Study IDs: ATR
Record Dates: First submitted 2024-03-30; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Cross Infection; Carbapenem Resistant Bacterial Infection; Vancomycin-Resistant Enterococcal Infection; Critical Illness
Keywords: Critical care; Healthcare Associated Infections; Drug resistance
MeSH Terms: conditions — Cross Infection; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- eHDR+: Patients with Emergent Highly Resistant Bacteria healthcare associated infection
  Interventions: Other: epidemiological records
- eHDR-: Patients without Emergent Highly Resistant Bacteria healthcare associated infection

INTERVENTIONS:
Other: epidemiological records — Healthcare associated infections due to emergent highly resistant bacteria, sites, risk factors, treatment and outcome
  Groups: eHDR+

SUMMARY:
Investigate the epidemiology, risk factors and impact on clinical practice of healthcare-associated infections with emergent highly drug-resistant (eHDR) pathogens, particularly carbapenem resistant enterobacteriaceae and glycopeptides-resistant enterococcus.

DETAILED DESCRIPTION:
In 2022, a previous one-day point-prevalence multicenter study (NOSOREA2, NCT05547646) showed that most prevalent pathogens causing healthcare-associated infections were carbapenem resistant enterobacteriaceae. In 2017, (NOSOREA1, LA TUNISIE MEDICALE - 2018 ; Vol 96 (10/11)), most prevalent pathogens were non-fermenting pathogens.

Faced with this major epidemiological change within Tunisian ICUs, we decided to launch a 3rd survey under the aegis of the 'Association tunisienne de réanimation'. We aimed to investigate the epidemiology, risk factors and impact on clinical practice of healthcare-associated infections with emergent highly drug-resistant (eHDR) pathogens, particularly carbapenem resistant enterobacteriaceae and glycopeptides-resistant enterococcus. So we conducted a multicenter prospective collection that will take place over 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients admitted during the study period

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients admitted during the study period
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Highly resistant bacterial healthcare associated infections | 2 months
  Incidence of eHRB healthcare associated infections in ICU
Epidemiological features of Highly resistant bacterial healthcare associated infections healthcare associated infections in ICU | 2 months
  Causative micro-organisms, sites and risk factors of eHRB healthcare associated infections in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Amira JAMOUSSI, Professor, Principal Investigator — Abderrahmen Mami Hospital
Locations (1):
- Abderrahmen Mami, Ariana, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided